CLINICAL TRIAL: NCT01318577
Title: Study of A New Contact Lens Cleaning and Disinfecting Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 682
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Vision Disorders
Keywords: Contact lens; Cleaning solution
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational Solution (Experimental): Hydrogen peroxide system for cleaning, protein removal, disinfecting and storing of contact lenses.
  Interventions: Device: Investigational Cleaning & Disinfecting Solution
- Clear Care Solution (Active Comparator): Hydrogen peroxide system for cleaning, protein removal, disinfecting and storing of contact lenses
  Interventions: Device: Clear Care Solution

INTERVENTIONS:
Device: Investigational Cleaning & Disinfecting Solution — Contact lenses will be cleaned and stored daily in the cleaning, disinfecting and storage solution
  Arms: Investigational Solution
Device: Clear Care Solution — Contact lenses will be cleaned and stored daily in the cleaning, disinfecting and storage solution
  Arms: Clear Care Solution

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of a new investigational cleaning and disinfecting solution (Test) compared to Clear Care cleaning and disinfecting solution (Control) when used by contact lens wearers to clean and disinfect their contact lenses for approximately three months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be habitual wearers of one of the protocol specified lenses.
* Subjects must habitually use a NON-PEROXIDE lens care product for cleaning, disinfecting and storage of their lenses.
* Subjects must be adapted lens wearers and wear a lens in each eye and each lens must be of the same manufacture and brand.
* Subjects must agree to wear their lenses on a daily wear basis for approximately three months.

Exclusion Criteria:

* Subjects who currently use a hydrogen peroxide cleaning and disinfecting solution.
* Subjects who currently wear Opaque Cosmetic Tint Contact Lenses.
* Subjects who have worn polymethylmethacrylate (PMMA) lenses within the last three months.
* Subjects with any systemic disease currently affecting ocular health or which in the Investigator"s opinion may have an effect on ocular health during the course of the study.
* Subjects using any systemic or topical medications that will, in the Investigator"s opinion, affect ocular physiology or lens performance.
* Subjects with any "Present" finding during the slit lamp examination that, in the Investigator"s judgment, interferes with contact lens wear.
* Subjects with any scar or neovascularization within the central 4 mm of the cornea.
* Subjects who are allergic to any component in the study care products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Barna, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Solution | Clear Care Solution
Started | 224 | 220
Completed | 211 | 212
Not Completed | 13 | 8

BASELINE CHARACTERISTICS:
Population: Demographics are reported for all eligible, dispensed subjects; 222 in the investigational group and 218 in the Clear Care group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Solution | Clear Care Solution | Total
Number analyzed (Participants) | 222 | 218 | 440
Age, Continuous [Mean (Full Range); unit: years] | 35.4 [18 to 68] | 35.3 [18 to 63] | 35.4 [18 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 163 | 323
  Male | 62 | 55 | 117

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With > Grade 2 Slit Lamp Findings
Description: Graded slit lamp findings for each eye, including epithelial edema, epithelial microcysts, corneal staining, limbal and bulbar injections, upper lid tarsal conjunctival abnormalities, corneal neovascularization, and corneal infiltrates were graded for severity on a scale from 0 (No Finding) to 4 (Severe Finding). The outcome measure is any finding > grade 2, across abnormalities.
Time Frame: 3 months
Population: There were 442 dispensed eyes with nonmissing scores in the investigational group and 438 dispensed eyes with nonmissing scores in the Clear Care group.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Investigational Solution | Clear Care Solution
Number analyzed (Participants) | 221 | 218
Number analyzed (eyes) | 442 | 436
eyes | 4 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events were not coded. Therefore, source vocabulary is not applicable. There were 448 eyes dispensed investigational solution and 440 eyes dispensed control solution, assessed for adverse events.
Arm/Group | Investigational Solution | Clear Care Solution
Serious Adverse Events (participants affected / at risk) | 0/224 | 0/220
Other Adverse Events (participants affected / at risk) | 0/224 | 0/220

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.